CLINICAL TRIAL: NCT01799863
Title: Artificial Tears Versus Preservative Free Ketorolac Trometamol 0.45% for Treatment of Acute Viral Conjunctivitis
Brief Title: Artificial Tears Versus Preservative Free Ketorolac Trometamol 0.45% for Acute Viral Conjunctivitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fundação Altino Ventura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAV011_12
Record Dates: First submitted 2013-02-22; First posted 2013-02-27 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Conjunctivitis, Viral
Keywords: Conjunctivitis, Viral; Ketorolac; Artificial tears
MeSH Terms: conditions — Conjunctivitis, Viral | interventions — Ketorolac; Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketorolac trometamol 0.45% (Experimental): Ketorolac trometamol 0.45% associated with carboxymethylcellulose eye drops (Acular CMC®, Allergan, Irvine, USA) qid for 7 days.
  Interventions: Drug: Ketorolac trometamol 0.45% with carboxymethylcellulose
- Artificial tears (Placebo Comparator): Preservative free artificial tears (Optive UD®, Allergan, Irvine, USA) qid for 7 days.
  Interventions: Drug: Preservative free artificial tear

INTERVENTIONS:
Drug: Ketorolac trometamol 0.45% with carboxymethylcellulose
  Other Names: Acular CMC®, Allergan, Irvine, USA
  Arms: Ketorolac trometamol 0.45%
Drug: Preservative free artificial tear
  Other Names: Optive UD®, Allergan, Irvine, USA
  Arms: Artificial tears

SUMMARY:
The purpose of this study is to evaluate the evolution of the symptoms of acute viral conjunctivitis using preservative free ketorolac trometamol 0.45% associated with carboxymethylcellulose compared with isolated use of preservative-free artificial tears.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the evolution of the symptoms of acute viral conjunctivitis using preservative free ketorolac trometamol 0.45% associated with carboxymethylcellulose compared with isolated use of preservative-free artificial tears. A randomized double-masked study will include 60 patients divided into two groups: Group 1: using a formulation of ketorolac tromethamine 0.45% associated with carboxymethylcellulose (Acular CMC®, Allergan, Irvine, USA) and Group 0: using artificial tears (Optive UD®, Allergan, Irvine, USA), both drugs without preservatives.

ELIGIBILITY:
Inclusion Criteria:

* Acute conjunctivitis (unilateral or bilateral) for less than two weeks,
* Signs and symptoms consistent with viral conjunctivitis and at least one of the following: preauricular lymphadenopathy, upper tract respiratory infection or recent contact with someone with conjunctivitis

Exclusion Criteria:

* pregnant women
* allergies to non-steroidal anti-inflammatories
* history of seasonal allergic conjunctivitis
* contact lens wearers
* history of ocular herpes infection
* blepharitis
* severe dry eye
* purulent discharge
* defects in the corneal epithelium

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in ocular symptoms from baseline to treatment day 7 | 7 days
  General ocular discomfort, itching, foreign body sensation, tearing, eye redness and eyelid edema. Symptoms will be graded as 0 (absence), I (mild), II (moderate) and III (severe).
Change in ocular signs from baseline to treatment day 7 | 7 days
  The clinical examination will consist of slit-lamp examination of the anterior segment. Four signs will be assessed: conjunctival hyperemia, chemosis, secretion and follicles in lower tarsal conjunctiva. The signs will be classified as 0 (absence), I (mild), II (moderate), III (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Falcão, MD, Principal Investigator — Fundação Altino Ventura; Lucio Maranhão, MD, Study Director — Fundação Altino Ventura
Locations (1):
- Fundação Altino Ventura, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Shiuey Y, Ambati BK, Adamis AP. A randomized, double-masked trial of topical ketorolac versus artificial tears for treatment of viral conjunctivitis. Ophthalmology. 2000 Aug;107(8):1512-7. doi: 10.1016/s0161-6420(00)00177-9. PMID 10919900
- [Background] Toker MI, Erdem H, Erdogan H, Arici MK, Topalkara A, Arslan OS, Pahsa A. The effects of topical ketorolac and indomethacin on measles conjunctivitis: randomized controlled trial. Am J Ophthalmol. 2006 May;141(5):902-905. doi: 10.1016/j.ajo.2005.12.004. Epub 2006 Mar 9. PMID 16527227